CLINICAL TRIAL: NCT03326440
Title: Virtual Environment Radiotherapy (VERT) to Improve Patients' Compliance to Radiotherapy (RT) in Prostate Cancer
Brief Title: Virtual Environment Radiotherapy to Improve Patients' Compliance to Radiotherapy (RT) in Prostate Cancer
Acronym: VERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 772
Record Dates: First submitted 2016-10-26; First posted 2017-10-31 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Arm (Other): Patients with a histological diagnosis of prostate cancer are shown how Radiotherapy is planned and given using 3D images on the VERT (Virtual Environment Radiotherapy) system prior to the start of Radiotherapy.
  Interventions: Other: VERT system
- Control Arm (Other): Patients with a histological diagnosis of prostate cancer who are shown how Radiotherapy is planned and given using 3D images on the VERT (Virtual Environment Radiotherapy) system following completion of Radiotherapy.
  Interventions: Other: VERT system

INTERVENTIONS:
Other: VERT system — 3D images of radiotherapy planning and administration using the VERT (Virtual Environment Radiotherapy) system is shown either prior to Radiotherapy (study arm) or post Radiotherapy (control arm)

SUMMARY:
Purpose of the study

1. To assess whether offering visual information to patients with prostate cancer prior to receiving RT increases the participant's compliance.
2. To assess whether increased compliance translates into reduced side effects from RT (assessed with a quality of life questionnaire).

Type of study. This is a randomised control trial which will include 170 patients with the histological diagnosis of prostate cancer in the study arm and 170 patients with the histological diagnosis of prostate cancer in the control/standard arm.

DETAILED DESCRIPTION:
The Oncology Department at the Royal Stoke University Hospital is a state of the art facility. It has radiotherapy (RT) facilities such as IMRT and rapid arc, leading the way in RT planning and delivery. The Investigators want to further their expertise and public involvement in RT planning with this proposal.

This study follows a pilot study in which patients receiving RT were shown how treatment is planned and given using a 3 dimensional (3D) imaging system. It was noticed that patients with prostate cancer entering the pilot study might have been more compliant (holding water before each treatment session) than those with prostate cancer not entering the study. On this basis, the investigators wish to run this project in which prostate cancer patients will be shown how RT is planned and given using 3D images prior to start RT (study arm, 170 patients) or after completion of RT (control/standard arm, 170 patients). A sample size calculation was performed (see below) in order to distinguish a 10% improvement in retention of bladder volume over the course of treatment.

RT planning will be carried out using standard procedures at the Oncology Department. However, each study patient's CT Scan image will be placed in the Virtual Environment for Radiotherapy Training (VERT) system. The original images will not be altered and will be presented using the established JImage Dicom libraries. 3D models will be constructed from the CT Images. The system allows moving the 3D images using a mouse. Planning CT Scans will be taken prior to RT, on the first 3 days, and once weekly during RT to measure bladder volumes (this is standard practice and no patients will have extra CT Scans). The investigators will assess whether patients in the study arm were more compliant in holding water when compared to control cases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the histological diagnosis of prostate cancer due to receive radical RT.
* Patients with prostate cancer deemed fit enough to complete a course of radical RT to their prostate area.
* Patients able to give informed consent.

Exclusion Criteria:

* The only exclusion criteria is for participants unable to understand the study aims and therefore unable to give informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-10-08; Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Volume of bladder measurement in cm3 | Through study completion, an average of seven and a half weeks.
  Measuring the bladder volume during Radiotherapy to assess if offering visual information to patients with prostate cancer prior to receiving radiotherapy increases their compliance.

SECONDARY OUTCOMES:
Does increased compliance translate into reduced side effects from RT. | Through study completion and follow up - an average of 8 months
  Data collection regarding radiotherapy side effects will be collected throughout the radiotherapy sessions and for 6 months after the radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Josep Sule-Suso, Principal Investigator — University Hospitals of North Midlands NHS Trust, Royal Stoke University Hospital, Oncology Department, City General Site, Newcastle Road, Stoke on Trent, ST4 6QG
Locations (1):
- University Hospitals of North Midlands, Royal Stoke University Hospital, City General Site, Newcaslte Road, Stoke-on-Trent, Staffordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No